CLINICAL TRIAL: NCT01690130
Title: Transcranial Magnetic Stimulation Effects on Nicotine Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Brain Stimulation Lab / MUSC
Record Dates: First submitted 2012-09-07; First posted 2012-09-21 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Nicotine Dependence
Keywords: nicotine; craving; smoking; TMS; prefrontal cortex
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Magnetic Stimulation (Experimental): Transcranial magnetic stimulation (TMS) is a noninvasive (and relatively painless) brain stimulation technology that can focally stimulate the brain of an awake individual.The brain stimulation techniques could theoretically improve the efficacy of smoking cessation. Treatment was standardized at 100% magnetic field intensity relative to the participant's resting MT, at 10 pulses per second (10 Hz) for 5 seconds, with an intertrain interval of 10 seconds. Treatment session lasted for 15 minutes with 3000 pulses.
  Interventions: Device: Transcranial Magnetic Stimulation (Neuronetics); Device: Sham Transcranial Magnetic Stimulation
- Sham Transcranial Magnetic Stimulation (Sham Comparator): Sham-TMS procedures: After rMT determination and DLPFC cortex localization, participants were fitted with two electrodes on the scalp just below the hairline. Electrodes were connected to an Epix VT® Transcutaneous Electrical Nerve Stimulation Device (Empi; St. Paul, MN, USA)
  Interventions: Device: Transcranial Magnetic Stimulation (Neuronetics); Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (Neuronetics) — Transcranial magnetic stimulation is a noninvasive brain stimulation that can focally stimulate the brain of an awake individual. A TMS pulse focally stimulates the cortex by depolarizing superficial neurons which induces electrical currents in the brain.
  Other Names: Neuronetics® Model 3600
Device: Sham Transcranial Magnetic Stimulation — The electrical current of the sham system is titrated to a level matching participants' ratings of active TMS.The sham-TMS scalp discomfort will be matched to that of active TMS.
  Other Names: Transcutaneous Electrical Nerve Stimulation Device

SUMMARY:
The proposed study will measure the change of cortical excitability during nicotine craving and examine the effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on nicotine craving and cue-reactivity among adult regular smokers.

DETAILED DESCRIPTION:
This pilot protocol proposes to test and further develop TMS for the purpose of studying brain function in nicotine users.

Specific Primary Aims include:

Aim # 1. To test change of cortical excitability during nicotine craving in cigarette smokers and explore the potential use of TMS in cigarette smokers.

Aim # 2. Given the role of the prefrontal cortex (and connected regions) in craving, we will examine whether modulating prefrontal activity through rTMS will impact measures of craving and the reinforcing effects of nicotine.

Design:

The study was a randomized, blind, sham-controlled crossover study in which participants will involve two study visits. Participants will have an initial assessment about tobacco use habits and craving patterns. Participant will look at images related to and not related to cigarette smoking.

Participants will receive two different types of brain stimulation with repetitive TMS (10 Hz): sham rTMS and active rTMS over prefrontal cortex. Craving assessments will be performed before and after each stimulus experiment.

Participants will be measured cortical excitability with TMS before and after each stimulus experiment.

ELIGIBILITY:
Inclusion Criteria:

* Right handed males and females, between the ages of 18 and 50
* Daily smokers who smoke at least 10 cigarettes per day for at least past 1 year
* Mentally capable of reading, writing, giving consent, following instructions

Exclusion Criteria:

* history of seizures
* taking medications that lower seizure threshold
* implanted metal devices (e.g., pacemakers, metal plates, wires)
* pregnant
* history of brain surgery or history of loss of consciousness >15 minutes
* any unstable major axis I psychiatric disorder in the past month (e.g. psychotic disorders)
* Current substance use disorders other than nicotine and caffeine use, in the past 30 days
* Any medication (e.g., propranolol) or unstable medical condition that may interfere with psychophysiological (e.g., heart rate) monitoring

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Amiaz R, Levy D, Vainiger D, Grunhaus L, Zangen A. Repeated high-frequency transcranial magnetic stimulation over the dorsolateral prefrontal cortex reduces cigarette craving and consumption. Addiction. 2009 Apr;104(4):653-60. doi: 10.1111/j.1360-0443.2008.02448.x. Epub 2009 Jan 12. PMID 19183128
- [Background] Eichhammer P, Johann M, Kharraz A, Binder H, Pittrow D, Wodarz N, Hajak G. High-frequency repetitive transcranial magnetic stimulation decreases cigarette smoking. J Clin Psychiatry. 2003 Aug;64(8):951-3. doi: 10.4088/jcp.v64n0815. PMID 12927012
- [Derived] Li X, Hartwell KJ, Owens M, Lematty T, Borckardt JJ, Hanlon CA, Brady KT, George MS. Repetitive transcranial magnetic stimulation of the dorsolateral prefrontal cortex reduces nicotine cue craving. Biol Psychiatry. 2013 Apr 15;73(8):714-20. doi: 10.1016/j.biopsych.2013.01.003. Epub 2013 Feb 26. PMID 23485014

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial Magnetic Stimulation, Then Sham: Transcranial magnetic stimulation (TMS) is a noninvasive (and relatively painless) brain stimulation technology that can focally stimulate the brain of an awake individual.The brain stimulation techniques could theoretically improve the efficacy of smoking cessation. Treatment was standardized at 100% magnetic field intensity relative to the participant's resting MT, at 10 pulses per second (10 Hz) for 5 seconds, with an intertrain interval of 10 seconds. Treatment session lasted for 15 minutes with 3000 pulses.
  Transcranial Magnetic Stimulation (Neuronetics): Transcranial magnetic stimulation is a noninvasive brain stimulation that can focally stimulate the brain of an awake individual. A TMS pulse focally stimulates the cortex by depolarizing superficial neurons which induces electrical currents in the brain.
- Sham Transcranial Magnetic Stimulation, Then TMS: Sham-TMS procedures: After rMT determination and DLPFC cortex localization, participants were fitted with two electrodes on the scalp just below the hairline. Electrodes were connected to an Epix VT® Transcutaneous Electrical Nerve Stimulation Device (Empi; St. Paul, MN, USA)
  Transcranial Magnetic Stimulation (Neuronetics): Transcranial magnetic stimulation is a noninvasive brain stimulation that can focally stimulate the brain of an awake individual. A TMS pulse focally stimulates the cortex by depolarizing superficial neurons which induces electrical currents in the brain.
  Sham Transcranial Magnetic Stimulation: The electrical current of the sham system is titrated to a level matching participants' ratings of active TMS.The sham-TMS scalp discomfort will be matched to that of active TMS.
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation, Then Sham | Sham Transcranial Magnetic Stimulation, Then TMS
Started | 10 | 9
Completed | 9 | 9
Not Completed | 1 | 0
Not completed — Subject have cancelled visit. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Magnetic Stimulation, Then Sham | Sham Transcranial Magnetic Stimulation, Then TMS | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 42 (11.5) | 42 (11.5) | 42 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: the Change From Baseline in Cue Nicotine Craving Rating Score
Description: Seventy highly palatable scenic images, forty neutral control images) and forty cigarette smoking cue images were presented in four blocks. Immediately after viewing each block of cue images, participants completed a 10 question computerized visual analog scale (CVAS) designed to assess craving. Each question is followed by a CVAS (range 0 - 100) 0 means least amount of craving and 100 means the maximum amount of craving. After 15 minutes of real or sham rTMS, participants viewed the images again and rated their cravings. At each visit, participants were blind to the rTMS condition (real or sham) and the order was randomized.
Time Frame: Before rMTS (baseline) and after rTMS experiment (on average 15 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 18 | 18
score on a scale | 64 (5.9) | 46 (6.4)

2. Secondary Outcome: the Change From Baseline in Resting Motor Threshold
Description: Resting Motor Threshold (RMT) on a scale from 0-100, with 100 being most power given to enact a motor response
Time Frame: 20 minutes before (baseline) and 20 minutes after rTMS experiment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 18 | 18
units on a scale | 42 (8.1) | 44 (9.8)

ADVERSE EVENTS:
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Magnetic Stimulation (N=19) | Sham Transcranial Magnetic Stimulation (N=19)
mild discomfort (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes